CLINICAL TRIAL: NCT02597933
Title: A Double Blind, Randomised, Placebo-controlled Trial Evaluating Efficacy and Safety of Oral Nintedanib Treatment for at Least 52 Weeks in Patients With Systemic Sclerosis Associated Interstitial Lung Disease (SSc-ILD)
Brief Title: A Trial to Compare Nintedanib With Placebo for Patients With Scleroderma Related Lung Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1199.214; 2015-000392-28 (EudraCT Number)
Record Dates: First submitted 2015-10-08; First posted 2015-11-05 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Scleroderma, Systemic
MeSH Terms: conditions — Scleroderma, Systemic | interventions — nintedanib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Nintedanib (Experimental): patient receives capsules containing nintedanib twice a day
  Interventions: Drug: Nintedanib
- Placebo (Placebo Comparator): patient receives capsules identical to those containing active drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nintedanib
  Arms: Nintedanib
Drug: Placebo
  Arms: Placebo

SUMMARY:
Systemic Sclerosis (SSc) is a devastating disease of unknown etiology. Patients suffer from multiple organ fibrosis whereas lung fibrosis (interstitial lung disease, ILD) is one of the main driver for mortality. There is preclinical evidence for efficacy of nintedanib in SSc and associated ILD (SSc-ILD) and the anti-fibrotic efficacy of nintedanib was proven in idiopathic pulmonary fibrosis patients, who are presenting a similar pattern regarding lung fibrosis. Hence it is the purpose of the trial to confirm the efficacy and safety of nintedanib 150 mg bid in treating patients with SSc-ILD, compared with placebo. The trial will be conducted as a double blind, randomised, placebo-controlled trial with primary efficacy evaluation at week 52 and placebo-controlled treatment until last patient out (up to a maximum of 100 weeks). Respiratory function is globally accepted for assessment of treatment effects in patients with lung fibrosis. The chosen endpoint (Forced Vital Capacity (FVC) decline) is easy to obtain and is part of the usual examinations done in patients with SSc-ILD.

ELIGIBILITY:
Inclusion criteria:

* Age >= 18 years
* 2013 American College of Rheumatology (ACR) / EULAR classification criteria for SSc fulfilled
* SSc disease onset (defined by first non-Raynaud symptom) within 7 years
* SSc related Interstitial Lung Disease confirmed by High Resolution Computer Tomography (HRCT); Extent of fibrotic disease in the lung >= 10%
* FVC >= 40% of predicted normal
* Carbon Monoxide Diffusion Capacity (DLCO) 30% to 89% of predicted normal

Exclusion criteria:

* Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) >1.5 x ULN
* Bilirubin >1.5 x ULN
* Creatinine clearance <30 mL/min
* Airway obstruction (pre-bronchodilator Forced Expiratory Volume in 1 second (FEV1)/FVC <0.7)
* Other clinically significant pulmonary abnormalities
* Significant Pulmonary Hypertension (PH)
* Cardiovascular diseases
* More than 3 digital fingertip ulcers or a history of severe digital necrosis requiring hospitalization or severe other ulcers
* Bleeding risk (such as predisposition to bleeding, fibrinolysis, full-dose anticoagulation, high dose antiplatelet therapy, history of hemorrhagic central nervous system (CNS) event within last year
* international normalised ratio (INR) >2, prolongation of prothrombin time (PT) and partial thromboplastin time (PTT) by >1.5 x ULN)
* History of thrombotic event within last year
* Clinical signs of malabsorption or needing parenteral nutrition
* Previous treatment with nintedanib or pirfenidone
* Treatment with prednisone >10 mg/day, azathioprine, hydroxychloroquine, colchicine, D-penicillamine, sulfasalazine, cyclophosphamide, rituximab, tocilizumab, abatacept, leflunomide, tacrolimus, newer anti-arthritic treatments like tofacitinib and cyclosporine A, potassium para-aminobenzoate
* Unstable background therapy with either mycophenolate mofetil or methotrexate
* Previous or planned hematopoietic stem cell transplantation
* Patients with underlying chronic liver disease (Child Pugh A, B, C hepatic impairment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (194):
- United States (44):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California Los Angeles, Los Angeles, California
  - University of California Davis, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - University of Florida College of Medicine, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic-Rochester, Rochester, Minnesota
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Hospital for Special Surgery, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center-New York Presbyterian Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Health, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Toledo, Toledo, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of South Carolina, Columbia, South Carolina
  - Vanderbilt Pulmonary Clinic, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University Of Texas at Houston, Houston, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (3):
  - Hospital Militar Central Cirujano Mayor Dr. Cosme Argerich, Buenos Aires
  - APRILLUS-Asistencia e Investigación, Ciudad Autonoma Buenos Aires
  - CEMER-Centro Medico De Enfermedades Respiratorias, Florida
- Australia (4):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
- Austria (2):
  - LKH-Univ. Hospital Graz, Graz
  - Medical University of Innsbruck, Innsbruck
- Belgium (5):
  - ULB Hopital Erasme, Brussels
  - Brussels - UNIV Saint-Luc, Brussels
  - UNIV UZ Gent, Ghent
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Edumed - Educacao e Saude SA, Curitiba, Brazil
- Canada (3):
  - Saint Joseph's Healthcare, Hamilton, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - HSCM, Montreal, Quebec
- Chile (2):
  - Hospital Clínico Reg. de Concepción "Dr. G. Grant Benavente", Concepción
  - Centro de Investigación del Maule, Talca
- China (9):
  - Peking Union Medical College Hospital, Beijing
  - Beijing Chao-Yang Hospital, Beijing
  - Beijing Hospital, Beijing
  - First Hospital of Jilin University, Changchun
  - West China Hospital, Chengdu
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Huashan Hospital, Fudan University, Shanghai
  - The First Hospital of Chinese Medical University, Shenyang
  - Zhuzhou Central Hospital, Zhuzhou
- Czechia (2):
  - Institute of Rheumathology Prague, Prague
  - Thomayer Hospital, Prague
- Denmark (2):
  - Aarhus Universitets Hospital, Aarhus
  - Odense Universitetshospital, Odense
- Finland (2):
  - HYKS Keuhkosairauksien, Helsinki
  - TYKS, Keuhkosairauksien klinikka, Turku, Turku
- France (13):
  - HOP Avicenne, Bobigny
  - HOP Louis Pradel, Bron
  - HOP Calmette, Lille
  - HOP Claude Huriez, Lille
  - HOP Arnaud de Villeneuve, Montpellier
  - HOP Hôtel-Dieu, Nantes
  - HOP Pasteur, Nice
  - HOP Cochin, Paris
  - HOP Bichat, Paris
  - HOP Pontchaillou, Rennes
  - HOP Charles Nicolle, Rouen
  - HOP Larrey, Toulouse
  - HOP Bretonneau, Tours
- Germany (13):
  - Kerckhoff-Klinik, Bad Nauheim, Bad Nauheim
  - Universitätsklinikum Köln (AöR), Cologne
  - Klinik Donaustauf, Donaustauf
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsmedizin Greifswald, Greifswald
  - Asklepios Klinik Altona, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Thoraxklinik-Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Klinikum der Universität München - Campus Großhadern, München
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Tübingen, Tübingen
- General Hospital of Athens "Laiko", Athens, Greece
- Semmelweis University, Dept. Pulmonology, Budapest, Hungary
- India (15):
  - St John's Medical College, Bangalore
  - Ramaiah Medical College and Hospitals, Bangalore
  - Mazumdar Shaw Medical centre, Bangalore
  - Postgraduate Institute of Medical Education And Research, Chandigarh
  - Care Hospital, Hyderabad
  - Nizam's Institute of Medical Sciences, Hyderabad
  - Asthma Bhawan, Jaipur
  - P.D. Hinduja National Hospital, Mumbai
  - Getwell Hospital & Research Institute, Nagpur
  - All India Institute of Medical Science, New Delhi
  - Sir Gangaram Hospital, New Delhi
  - Jehangir Clinical Development Centre Pvt. Ltd., Pune
  - B.J. Medical College and Sasoon General Hospital, Pune
  - Inamdar Multispeciality Hospital, Pune
  - Christian Medical College, Vellore
- Ireland (2):
  - Cork University Hospital, Cork
  - Mater Misericordiae University Hospital, Dublin
- Israel (4):
  - Bnei Zion Medical Center, Haifa, Haifa
  - Rambam Medical Center, Haifa
  - Rabin Medical Center Beilinson, Petah Tikva
  - Sourasky Medical Center, Tel Aviv
- Italy (6):
  - Az. Ospedaliere Umberto I di Ancona, Ancona
  - Università degli Studi di Genova, Genova
  - A.O. San Gerardo di Monza, Monza
  - A.O Universitaria - Università degli Studi della Campania Luigi Vanvitelli, Napoli
  - Università degli Studi Padova, Padua
  - Azienda Universitaria-Universita' La Sapienza, Roma
- Japan (20):
  - Tosei General Hospital, Aichi, Seto
  - Kurume University Hospital, Fukuoka, Kurume
  - Sapporo Medical University Hospital, Hokkaido, Sapporo
  - National Hospital Organization Himeji Medical Center, Hyogo, Himeji
  - Iwate Medical University Hospital, Iwate, Morioka
  - St. Marianna University School of Medicine Hospital, Kanagawa, Kawasaki
  - Kitasato University Hospital, Kanagawa, Sagamihara
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - Kyoto University Hospital, Kyoto, Kyoto
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Kindai University Hospital, Osaka, Osakasayama
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Osaka, Sakai
  - Osaka Medical College Hospital, Osaka, Takatsuki
  - Saitama Medical University Hospital, Saitama, Iruma-gun
  - Hamamatsu University Hospital, Shizuoka, Hamamatsu
  - Tokushima University Hospital, Tokushima, Tokushima
  - Juntendo University Hospital, Tokyo, Bunkyo-Ku
  - Nippon Medical School Hospital, Tokyo, Bunkyo-Ku
  - Toho University Omori Medical Center, Tokyo, Ota-ku
  - Institute of Rheumatology Tokyo Women's Medical University, Tokyo, Shinjyuku-ku
- Malaysia (4):
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Selayang, Kuala Selangor
  - Hospital Pulau Pinang, Pulau Pinang
  - Hospital Tuanku Ja'afar, Seremban
- Instituto Nacional de Enfermedades Respiratorias Ismael Cosío Villegas, Mexico City, Mexico
- Netherlands (4):
  - VU Medisch Centrum, Amsterdam
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - Radboud Universitair Medisch Centrum, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
- Norway (2):
  - Oslo Universitetssykehus HF, Rikshospitalet, Oslo
  - Universitetssykehuset Nord-Norge, Tromsø, Tromsø
- Poland (4):
  - Dr.Biziel UnivHosp#2,Rheumat&Connec.Tissue Disease,Bydgoszcz, Bydgoszcz
  - Dobry Lekarz,Spec.Med.Clinics,Private Prac,Krakow, Krakow
  - EMED, Center of Medical Services,Private Prac,Rzeszow, Rzeszów
  - Indep.Pblic Clin.Hosp#1,Dermatol,Venereol&Allerg.dep,Wroclaw, Wroclaw
- Portugal (6):
  - Hospital Garcia de Orta, EPE, Almada
  - Hospital Fernando Fonseca, EPE, Amadora
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - ULSAM, EPE - Hospital Conde de Bertiandos, Ponte de Lima
  - Centro Hospitalar São João,EPE, Porto
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia
- Spain (8):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Dr. Peset, Valencia
  - Hospital Politècnic La Fe, Valencia
  - Hospital Álvaro Cunqueiro, Vigo
- Clinical Rheumatology Research Center Sahlgrenska, Gothenburg, Sweden
- Switzerland (2):
  - Kantonspital St. Gallen, Rheumatologie Department, Sankt Gallen
  - Universitätsspital Zürich, Zurich
- Thailand (3):
  - Songklanagarind Hospital, Hat Yai
  - Srinagarind Hospital, Muang
  - Ramathibodi Hospital, Ratchathewi
- United Kingdom (5):
  - Glasgow Royal Infirmary, Glasgow
  - Royal Free Hospital, London
  - Guy's Hospital, London
  - Royal Brompton Hospital, London
  - Salford Royal Hospital, Salford

REFERENCES:
- [Derived] Volkmann ER, Assassi S, Denton CP, Simonovska R, Sambevski S, Alves M, Bernstein EJ. Outcomes in Systemic Sclerosis-Associated Interstitial Lung Disease Based on Serological Profiles With a Focus on Anticentromere and Anti-RNA Polymerase III Antibodies. J Rheumatol. 2025 Sep 1;52(9):914-918. doi: 10.3899/jrheum.2024-1063. PMID 40233987
- [Derived] Volkmann ER, McMahan ZH, Smith V, Jouneau S, Miede C, Alves M, Herrick AL; SENSCIS Trial Investigators. Risk of Malnutrition in Patients With Systemic Sclerosis-Associated Interstitial Lung Disease Treated With Nintedanib in the Randomized, Placebo-Controlled SENSCIS Trial. Arthritis Care Res (Hoboken). 2023 Dec;75(12):2501-2507. doi: 10.1002/acr.25176. Epub 2023 Aug 7. PMID 37357024
- [Derived] Allanore Y, Khanna D, Smith V, Aringer M, Hoffmann-Vold AM, Kuwana M, Merkel PA, Stock C, Sambevski S, Denton CP; SENSCIS Trial Investigators. Effects of nintedanib in patients with limited cutaneous systemic sclerosis and interstitial lung disease. Rheumatology (Oxford). 2024 Mar 1;63(3):639-647. doi: 10.1093/rheumatology/kead280. PMID 37294870
- [Derived] Denton CP, Goh NS, Humphries SM, Maher TM, Spiera R, Devaraj A, Ho L, Stock C, Erhardt E, Alves M, Wells AU. Extent of fibrosis and lung function decline in patients with systemic sclerosis and interstitial lung disease: data from the SENSCIS trial. Rheumatology (Oxford). 2023 May 2;62(5):1870-1876. doi: 10.1093/rheumatology/keac535. PMID 36111858
- [Derived] Maher TM, Bourdin A, Volkmann ER, Vettori S, Distler JHW, Alves M, Stock C, Distler O. Decline in forced vital capacity in subjects with systemic sclerosis-associated interstitial lung disease in the SENSCIS trial compared with healthy reference subjects. Respir Res. 2022 Jul 5;23(1):178. doi: 10.1186/s12931-022-02095-6. PMID 35790961
- [Derived] Kreuter M, Hoffmann-Vold AM, Matucci-Cerinic M, Saketkoo LA, Highland KB, Wilson H, Alves M, Erhardt E, Schoof N, Maher TM. Impact of lung function and baseline clinical characteristics on patient-reported outcome measures in systemic sclerosis-associated interstitial lung disease. Rheumatology (Oxford). 2023 Feb 6;62(SI):SI43-SI53. doi: 10.1093/rheumatology/keac325. PMID 35640959
- [Derived] Volkmann ER, Kreuter M, Hoffmann-Vold AM, Wijsenbeek M, Smith V, Khanna D, Denton CP, Wuyts WA, Miede C, Alves M, Sambevski S, Allanore Y. Dyspnoea and cough in patients with systemic sclerosis-associated interstitial lung disease in the SENSCIS trial. Rheumatology (Oxford). 2022 Nov 2;61(11):4397-4408. doi: 10.1093/rheumatology/keac091. PMID 35150246
- [Derived] Kreuter M, Del Galdo F, Miede C, Khanna D, Wuyts WA, Hummers LK, Alves M, Schoof N, Stock C, Allanore Y. Impact of lung function decline on time to hospitalisation events in systemic sclerosis-associated interstitial lung disease (SSc-ILD): a joint model analysis. Arthritis Res Ther. 2022 Jan 10;24(1):19. doi: 10.1186/s13075-021-02710-9. PMID 35012623
- [Derived] Highland KB, Distler O, Kuwana M, Allanore Y, Assassi S, Azuma A, Bourdin A, Denton CP, Distler JHW, Hoffmann-Vold AM, Khanna D, Mayes MD, Raghu G, Vonk MC, Gahlemann M, Clerisme-Beaty E, Girard M, Stowasser S, Zoz D, Maher TM; SENSCIS trial investigators. Efficacy and safety of nintedanib in patients with systemic sclerosis-associated interstitial lung disease treated with mycophenolate: a subgroup analysis of the SENSCIS trial. Lancet Respir Med. 2021 Jan;9(1):96-106. doi: 10.1016/S2213-2600(20)30330-1. PMID 33412120
- [Derived] Roennow A, Sauve M, Welling J, Riggs RJ, Kennedy AT, Galetti I, Brown E, Leite C, Gonzalez A, Portales Guiraud AP, Houyez F, Camp R, Gilbert A, Gahlemann M, Moros L, Luna Flores JL, Schmidt F, Sauter W, Finnern H. Collaboration between patient organisations and a clinical research sponsor in a rare disease condition: learnings from a community advisory board and best practice for future collaborations. BMJ Open. 2020 Dec 16;10(12):e039473. doi: 10.1136/bmjopen-2020-039473. PMID 33328257
- [Derived] Azuma A, Chung L, Behera D, Chung M, Kondoh Y, Ogura T, Okamoto M, Swarnakar R, Zeng X, Zou H, Meng X, Gahlemann M, Alves M, Kuwana M; SENSCIS trial investigators. Efficacy and safety of nintedanib in Asian patients with systemic sclerosis-associated interstitial lung disease: Subgroup analysis of the SENSCIS trial. Respir Investig. 2021 Mar;59(2):252-259. doi: 10.1016/j.resinv.2020.10.005. Epub 2020 Nov 19. PMID 33223487
- [Derived] Maher TM, Mayes MD, Kreuter M, Volkmann ER, Aringer M, Castellvi I, Cutolo M, Stock C, Schoof N, Alves M, Raghu G; SENSCIS Trial Investigators. Effect of Nintedanib on Lung Function in Patients With Systemic Sclerosis-Associated Interstitial Lung Disease: Further Analyses of a Randomized, Double-Blind, Placebo-Controlled Trial. Arthritis Rheumatol. 2021 Apr;73(4):671-676. doi: 10.1002/art.41576. Epub 2021 Mar 8. PMID 33142016
- [Derived] Kuwana M, Ogura T, Makino S, Homma S, Kondoh Y, Saito A, Ugai H, Gahlemann M, Takehara K, Azuma A. Nintedanib in patients with systemic sclerosis-associated interstitial lung disease: A Japanese population analysis of the SENSCIS trial. Mod Rheumatol. 2021 Jan;31(1):141-150. doi: 10.1080/14397595.2020.1751402. Epub 2020 Apr 23. PMID 32243207
- [Derived] Distler O, Highland KB, Gahlemann M, Azuma A, Fischer A, Mayes MD, Raghu G, Sauter W, Girard M, Alves M, Clerisme-Beaty E, Stowasser S, Tetzlaff K, Kuwana M, Maher TM; SENSCIS Trial Investigators. Nintedanib for Systemic Sclerosis-Associated Interstitial Lung Disease. N Engl J Med. 2019 Jun 27;380(26):2518-2528. doi: 10.1056/NEJMoa1903076. Epub 2019 May 20. PMID 31112379
- [Derived] Distler O, Brown KK, Distler JHW, Assassi S, Maher TM, Cottin V, Varga J, Coeck C, Gahlemann M, Sauter W, Schmidt H, Highland KB; SENSCIS trial investigators. Design of a randomised, placebo-controlled clinical trial of nintedanib in patients with systemic sclerosis-associated interstitial lung disease (SENSCIS). Clin Exp Rheumatol. 2017 Sep-Oct;35 Suppl 106(4):75-81. Epub 2017 Jun 29. PMID 28664834

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, placebo-controlled, double-blind, parallel design trial.
  Abbreviation used:
  treatment (trt) baseline (bl.) categorical (cat.) continuous (cont.) number (no.) patient (pt) Placebo (pl.) discontinued (disc.) primary analysis (PA) Antitopoisomerase Antibody (ATA)
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist sites to ensure that they (the subjects) met all implemented inclusion/exclusion criteria. Subjects were not to be randomised to trial drug if any of the specific entry criteria was violated
Groups:
- Placebo: Patients were administered orally placebo matching nintedanib 150 milligram (mg) soft gelatine capsules, twice daily with a possibility to interrupt treatment or to reduce to 100mg to manage adverse events.
- Nintedanib: Patients were administered orally 150 milligram (mg) soft gelatin capsules, twice daily with a possibility to interrupt treatment or to reduce to 100mg to manage adverse events.
Period: Overall Study
Arm/Group | Placebo | Nintedanib
Started | 290 (Started are randomised) | 290 (Started are randomised)
Treated Patients | 288 | 288
Completed | 252 | 239
Not Completed | 38 | 51
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Protocol Violation | 2 | 2
Not completed — Adverse Event | 20 | 28
Not completed — Not treated | 2 | 2
Not completed — Other than stated above | 7 | 14

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set consisted of patients who were randomised to a treatment group and received at least 1 dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nintedanib | Total
Number analyzed (Participants) | 288 | 288 | 576
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.4 (12.6) | 54.6 (11.8) | 54.0 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 221 | 433
  Male | 76 | 67 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 22 | 40
  Not Hispanic or Latino | 270 | 266 | 536
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 81 | 62 | 143
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 16 | 20 | 36
  White | 186 | 201 | 387
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Baseline pulmonary efficacy variables - Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: mL] | 2541.0 (815.5) | 2458.5 (735.9) | 2499.7 (777.2)

OUTCOME MEASURES:

1. Primary Outcome: Annual Rate of Decline in Forced Vital Capacity (FVC) Over 52 Weeks
Description: Forced vital capacity (FVC) is the total amount of air exhaled during the lung function test.
  For this endpoint reported means represent the adjusted rate.
Time Frame: up to week (wk) 52 after the start of administration
Population: Treated Set
Measure: Mean (Standard Error); unit: millilitre (mL)/year (yr)
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 288 | 288
millilitre (mL)/year (yr) | -93.3 (13.5) | -52.4 (13.8)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib; The primary analysis is a restricted maximum likelihood (REML) based approach using a random slope & intercept model. The analysis included the fixed, categorical effects of treatment, ATA status & gender, fixed continuous effects of time & baseline FVC (mL), age and height as well as the treatment-by time & baseline-by-time interactions. Random effects was included for patient response for both time & intercept.Within-patient errors are modelled by an unstructured variance-covariance matrix; Test type: Other; p = 0.0350, random coefficient regression; Mean Difference (Final Values) = 40.95, 95% CI 2-sided [2.88 to 79.01], Standard Error of Mean 19.38 — The model assumed that data were missing at random & that patients who dropped out would have behaved similarly to those who remained in trial
Statistical Analysis 2: Comparison: Placebo vs Nintedanib; This is a sensitivity analysis (SA) on primary endpoint including only on-trt measurements of FVC [mL]. The random coefficient model was used. The analysis included fixed, categorical effects of trt, ATA status & gender, fixed continuous effects of time & bl. FVC (mL), age, height, trt -by time & bl.-by-time interactions. Random effects included for patient response for both time & intercept. Within-patient errors were modelled by an Unstructured variance-covariance matrix; Test type: Other; p = 0.0378, random coefficient regression; The model assumed that data were missing at random & that patients who dropped out would have behaved similarly to those who remained in trial; Mean Difference (Final Values) = 43.13, 95% CI 2-sided [2.44 to 83.83]
Statistical Analysis 3: Comparison: Placebo vs Nintedanib; In multiple imputation SA 1, missing FVC values at wk 52 in pts who were alive at wk 52 were imputed assuming similar rate of FVC decline as in pts from corresponding trt group who prematurely disc. trial drug but had wk 52 FVC value. Missing FVC values at wk 52 in pts who died before wk 52 were imputed assuming similar rate of FVC decline as in pl. pts with wk 52 FVC value who prematurely disc. trial drug with most severe declines.The imputation model was similar to statistical model of PA; Test type: Other; p = 0.1046, random coefficient regression; Mean Difference (Final Values) = 30.00, 95% CI 2-sided [-6.22 to 66.22]
Statistical Analysis 4: Comparison: Placebo vs Nintedanib; In multiple imputation SA 2, missing FVC values at wk 52 in pts who were alive at wk 52 were imputed assuming similar rate of FVC decline as in pts from pl. group who prematurely disc. trial drug but had a wk 52 FVC value. Missing FVC values at wk 52 in pts who died before wk 52 were imputed assuming similar rate of FVC decline as in pl. pts with a wk 52 FVC value who prematurely disc. trial drug with most severe declines. The imputation model was similar to the statistical model of the PA; Test type: Other; p = 0.0740, random coefficient regression; Mean Difference (Final Values) = 32.93, 95% CI 2-sided [-3.19 to 69.06]
Statistical Analysis 5: Comparison: Placebo vs Nintedanib; In multiple imputation SA 3, missing FVC values at wk 52 in pts who were alive at wk 52 were imputed assuming a similar rate of FVC decline as in all pts in the pl. group who were included in the PA. Missing FVC values at wk 52 in pts who died before wk 52 were imputed assuming a similar rate of FVC decline as in all placebo patients included in the primary analysis with the most severe declines. The imputation model was similar to the statistical model of the PA; Test type: Other; p = 0.0644, random coefficient regression; Mean Difference (Final Values) = 33.86, 95% CI 2-sided [-2.03 to 69.75]
Statistical Analysis 6: Comparison: Placebo vs Nintedanib; This is sensitivity analysis using the model similar to the primary analysis but including a different set of covariates: the fixed, categorical effects of treatment, ATA status, the fixed continuous effects of time, baseline FVC (mL), and the treatment-by-time and baseline-by-time interactions.Random effects was included for patient response for both time and intercept; Test type: Other; p = 0.0351, random coefficient regression; Mean Difference (Final Values) = 40.95, 95% CI 2-sided [2.88 to 79.01]
Statistical Analysis 7: Comparison: Placebo vs Nintedanib; This is sensitivity analysis using the model similar to the primary analysis but including a different set of covariates: the fixed, categorical effects of treatment, ATA status (Positive / Negative), gender and mycophenolate mofetil /sodium background therapy use (Yes / No), fixed continuous effects of time, age , height and baseline FVC (mL), the treatment-by-time and baseline-by-time interactions. Random effects was included for patient response for both time and intercept; Test type: Other; p = 0.0349, random coefficient regression; Mean Difference (Final Values) = 40.98, 95% CI 2-sided [2.92 to 79.04]

2. Secondary Outcome: Absolute Change From Baseline in the Modified Rodnan Skin Score (mRSS) at Week 52
Description: This is the first key secondary endpoint.
  The modified Rodnan Skin Score (mRSS) is an evaluation of the patient's skin thickness rated by clinical palpation using a 0 to 3 scale. The scale differentiates between 0 = normal skin, 1 = mild thickness, 2 = moderate thickness, and 3 = severe thickness with inability to pinch the skin into a fold.
  The palpation is done for each of the 17 surface anatomic areas of the body: face, anterior chest, abdomen, fingers (right and left separately), forearms, upper arms, thighs, lower legs, dorsum of hands and feet. The sum of these individual values is defined as the total skin score. The mRSS has a range from 0 (no thickening) to 51 (severe thickening in all 17 areas). A high score corresponds to worse skin thickness.
  Least square mean is actually the adjusted mean. Adjusted mean was based on all analysed patients in the model (not only patients with a baseline and measurement at Week 52).
Time Frame: Baseline and up to 52 weeks after the start of administration
Population: Treated Set
Measure: Least Squares Mean (Standard Error); unit: unit on scale
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 288 | 288
unit on scale | -1.96 (0.26) | -2.17 (0.27)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib; The mixed model repeated measures (MMRM) approach was used. The model assumed that data were missing at random & that patients who dropped out would have behaved similarly to those who remained in trial; Test type: Other; p = 0.5785, MMRM; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.94 to 0.53], Standard Error of Mean 0.37

3. Secondary Outcome: Absolute Change From Baseline in Saint George's Respiratory Questionnaire (SGRQ) Total Score at Week 52.
Description: This is the second key secondary endpoint.
  The Saint George's Respiratory Questionnaire measures the health status in patients with chronic airflow limitation. It consists of 2 parts that cover 3 domains: symptoms, activities, and impacts. The symptom domain relates to the effect, frequency and severity of respiratory symptoms. The activity domain relates to activities that cause or are limited by breathlessness. The impact domain evaluates a range of aspects concerned with social functioning and psychological disturbances resulting from airways disease. The scores of these domains range from 0 (no impairment) to 100 (worst possible). The calculated total score summarises the impact of the disease on overall health status. A high score corresponds to worse health.
  Least square mean is actually the adjusted mean. Adjusted mean was based on all analysed patients in the model (not only patients with a baseline and measurement at Week 52).
Time Frame: Baseline and up to 52 weeks after the start of administration
Population: Treated set
Measure: Least Squares Mean (Standard Error); unit: unit on scale
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 288 | 288
unit on scale | -0.88 (0.87) | 0.81 (0.88)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib; Based on mixed model repeated measures (MMRM) approach was used, with fixed categorical effects of ATA status, visit, treatment-by visit interaction and baseline-by-visit interaction. Visit was the repeated measure. Within-patient errors were modelled by unstructured variance-covariance structure; Test type: Other; p = 0.1711, MMRM; The MMRM model assumed that data were missing at random & that patients who dropped out would have behaved similarly to those who remained in trial; Mean Difference (Final Values) = 1.69, 95% CI 2-sided [-0.73 to 4.12], Standard Error of Mean 1.24

4. Secondary Outcome: Annual Rate of Decline in FVC in Percentage (%) Predicted Over 52 Weeks
Description: Annual rate of decline in FVC in percentage (%) predicted over 52 weeks.
  For this endpoint reported means represent the adjusted rate.
Time Frame: up to 52 weeks after the start of administration
Population: Treated set
Measure: Mean (Standard Error); unit: % predicted/yr
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 288 | 288
% predicted/yr | -2.6 (0.4) | -1.4 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib; Based on a random coefficient regression with fixed categorical effects of treatment, ATA status, fixed continuous effects of time, baseline FVC [% pred], & including treatment-by-time and baseline-by-time interactions. Random effect was included for patient specific intercept & time. Within-patient errors are modelled by an Unstructured variance-covariance matrix. Inter-individual variability is modelled by a Variance-Components variance-covariance matrix; Test type: Other; p = 0.0331, MMRM; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = 1.15, 1.15% CI 2-sided [0.09 to 2.21], Standard Error of Mean 0.54

5. Secondary Outcome: Absolute Change From Baseline in FVC in mL at Week 52
Description: Absolute change from baseline in FVC in mL at Week 52. Least square mean is actually the adjusted mean. Adjusted mean was based on all analysed patients in the model (not only patients with a baseline and measurement at Week 52).
Time Frame: Baseline and up to 52 weeks after the start of administration
Population: Treated Set
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 288 | 288
mL | -101.03 (13.62) | -54.63 (13.94)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib; Based on mixed model repeated measures (MMRM) approach was used, with fixed categorical effects of ATA status, visit, treatment-by-visit interaction and baseline-by-visit interaction. Visit was the repeated measure. Within-patient errors were modelled by unstructured variance-covariance structure; Test type: Other; p = 0.0177, MMRM; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = 46.41, 95% CI 2-sided [8.09 to 84.73], Standard Error of Mean 19.51

6. Secondary Outcome: Relative Change From Baseline [%] of mRSS at Week 52
Description: Relative change from baseline [%] of mRSS at Week 52.
  The modified Rodnan Skin Score (mRSS) is an evaluation of the patient's skin thickness rated by clinical palpation using a 0 to 3 scale. The scale differentiates between 0 = normal skin, 1 = mild thickness, 2 = moderate thickness, and 3 = severe thickness with inability to pinch the skin into a fold.
  The palpation is done for each of the 17 surface anatomic areas of the body: face, anterior chest, abdomen, fingers (right and left separately), forearms, upper arms, thighs, lower legs, dorsum of hands and feet. The sum of these individual values is defined as the total skin score. The mRSS has a range from 0 (no thickening) to 51 (severe thickening in all 17 areas). A high score corresponds to worse skin thickness.
  Least square mean is actually the adjusted mean. Adjusted mean was based on all analysed patients in the model (not only patients with a baseline and measurement at Week 52).
Time Frame: Baseline and up to 52 weeks after the start of administration
Population: Treated set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 288 | 288
percent change | -3.92 (5.89) | -10.20 (5.98)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.4547, MMRM; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = -6.28, 95% CI 2-sided [-22.77 to 10.21], Standard Error of Mean 8.39

7. Secondary Outcome: Time to Death
Description: Time to event analysis of patients with death. The number of observed patients with death are reported.
Time Frame: From date of first trial drug intake up to date of death or last contact date (ie., up to 100 weeks)
Population: Treated set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 288 | 288
Participants | 9 | 10
Statistical Analysis 1: Comparison: Placebo vs Nintedanib; Test type: Other; p = 0.7535, Regression, Cox; Based on Cox's regression model (Wald test), stratified by ATA status; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.47 to 2.84]

8. Secondary Outcome: The Percentage (%) of Responder Based on Combined Response Index in Systemic Sclerosis (CRISS) at Week 52
Description: The percentage (%) of responder based on Combined Response Index in Systemic Sclerosis (CRISS) at Week 52.
  This is a composite endpoint, based on the mRSS, FVC percent predicted, HAQ-DI, patient's global impression of overall health Visual Analogue Scale (VAS) and physician's global impression of patient's overall health VAS, as well as the absence of significant worsening of interstitial lung disease, a new scleroderma renal crisis, left ventricular failure or pulmonary arterial hypertension.
  The CRISS index score represents a probability of improvement and ranges between 0 and 1.
  This is a 2 stage process to predict probability of improvement:
  Step 1 - absence of major organ progression (SRC etc.) - score "0" Step 2 - predicted probability of improvement - (score "0 - 1")
Time Frame: Week 52
Population: Treated set
Measure: Number; unit: (%) of responder based on CRISS
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 288 | 288
(%) of responder based on CRISS | 11.8 | 12.2
Statistical Analysis 1: Comparison: Placebo vs Nintedanib; The comparison between both treatment groups was performed using a Cochran-Mantel-Haenszel test. CRISS score at Week 52 was transformed into 100 binary responder endpoints using multiple imputation. These were analyzed using a Cochran-Mantel-Haenszel test, stratified by ATA status OR and the 95% confidence interval (CI) as obtained from all 100 imputations were combined using Rubin´s rule; Test type: Other; p = 0.9115, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.57 to 1.88]; Missing values were imputed using worst case, i.e. considered having disease progression

9. Secondary Outcome: Absolute Change From Baseline in Carbon Monoxide Diffusion Capacity (DLco) in % Predicted at Week 52
Description: Absolute change from baseline in Carbon Monoxide Diffusion Capacity (DLco) in % predicted at Week 52.
  Least square mean is actually the adjusted mean. Adjusted mean is based on all analysed patients in the model (not only patients with a baseline and measurement at week 52).
Time Frame: Baseline and up to 52 weeks after the start of administration
Population: Treated set
Measure: Least Squares Mean (Standard Error); unit: % predicted DLco
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 288 | 288
% predicted DLco | -2.77 (0.54) | -3.21 (0.54)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.5668, MMRM; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-1.94 to 1.06], Standard Error of Mean 0.76

10. Secondary Outcome: Absolute Change From Baseline in Digital Ulcer Net Burden at Week 52
Description: Absolute change from baseline in digital ulcer net burden (defined as the number of new digital ulcers (DUs) plus the number of DUs that have been verified at any earlier assessment during the trial) at Week 52.
  It is calculated at a visit by counting the total number of fingertips with ulcers (i.e. number of fingers with presence of digital ulcer ticked "Yes") at the corresponding visit
  Least square mean is actually the adjusted mean. Adjusted mean is based on all analysed patients in the model (not only patients with a baseline and measurement at week 52).
Time Frame: Baseline and up to 52 weeks after the start of administration
Population: Treated set
Measure: Least Squares Mean (Standard Error); unit: fingers
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 288 | 288
fingers | 0.06 (0.04) | 0.03 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.5914, MMRM; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.16 to 0.09], Standard Error of Mean 0.06

11. Secondary Outcome: Absolute Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 52
Description: Absolute change from baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) score at Week 52.
  The HAQ-DI score is calculated as follows:
  Each question is scored 0-3 (where 0= "without difficulty" & 3= "unable to do"). There are 8 categories (Dressing & Grooming, Arising, Eating, Walking, Hygiene, Reach, Grip, Activities), each including 2 or 3 questions. The score for each category corresponds to maximum question score within each category.
  Finally, HAQ-DI score corresponds to sum of the sub-scores of all 8 categories divided by number of categories completed. Please note that if there are fewer than 6 categories with responses, then a score cannot be calculated.
  The HAQ-DI score scale has 25 possible values (i.e., 0, 0.125, 0.250, 0.375 … 3). A high score corresponds to worse impairment.
  Least square mean is actually the adjusted mean. Adjusted mean is based on all analysed patients in the model (not only patients with a baseline and measurement at week 52).
Time Frame: Baseline and up to 52 weeks after the start of administration
Population: Treated set
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 288 | 288
unit on a scale | 0.022 (0.024) | 0.054 (0.024)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.3447, MMRM; Mean Difference (Final Values) = 0.032, 95% CI 2-sided [-0.035 to 0.099], Standard Error of Mean 0.034

12. Secondary Outcome: Absolute Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT) Dyspnoea Score at Week 52
Description: Absolute change from baseline in Functional Assessment of Chronic Illness Therapy (FACIT) dyspnoea score at Week 52.
  FACIT-Dyspnoea (Dyspnoea) 10 Item Short Form include a 4-point rating scale (no shortness of breath=0; mildly short of breath=1; moderately short of breath = 2; severely short of breath =3; or I did not do this in the past 7 days =4).
  A raw score is calculated as: Sum individual item scores * 10 / number of items answered. Raw scores are then converted to scale scores using the table included in the FACIT Dyspnoea Scale Short Form Scoring Guideline. FACIT dyspnea scale score ranges between 0 and 75.9.
  The FACIT-Dyspnea short forms are scored such that a high score represents high levels of dyspnea.
  Least square mean is actually the adjusted mean. Adjusted mean is based on all analysed patients in the model (not only patients with a baseline and measurement at week 52).
Time Frame: Baseline and up to 52 weeks after the start of administration
Population: Treated set
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 288 | 288
Unit on a scale | 0.34 (0.41) | 0.99 (0.42)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.2727, MMRM; Mean Difference (Final Values) = 0.64, 95% CI 2-sided [-0.51 to 1.79], Standard Error of Mean 0.58

ADVERSE EVENTS:
Time Frame: From date of first trial drug intake up to date of death or last contact date (ie., up to 100 weeks)
Arm/Group | Placebo | Nintedanib
All-Cause Mortality (participants affected / at risk) | 9/288 | 10/288
Serious Adverse Events (participants affected / at risk) | 79/288 | 88/288
Other Adverse Events (participants affected / at risk) | 239/288 | 270/288
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=288) | Nintedanib (N=288)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 3 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 1
Pleuropericarditis (Cardiac disorders) | 0 | 1
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 1
Macular oedema (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Retinal vein occlusion (Eye disorders) | 1 | 0
Rhegmatogenous retinal detachment (Eye disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Intestinal mass (Gastrointestinal disorders) | 1 | 0
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Brain death (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Polyp (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 1
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 1
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 | 2
Adenovirus infection (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 2
Gangrene (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 2
Lung infection (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 10
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 3
Sepsis (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Systemic candida (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Cell marker increased (Investigations) | 1 | 0
Forced vital capacity decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Drooping shoulder syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic scleroderma (Musculoskeletal and connective tissue disorders) | 2 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Sweat gland tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery aneurysm (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebral amyloid angiopathy (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral microhaemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 3
Bladder perforation (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Scleroderma renal crisis (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 3
Vulvovaginal swelling (Reproductive system and breast disorders) | 1 | 0
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 6 | 10
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Systemic sclerosis pulmonary (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Digital pitting scar (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Sclerema (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Raynaud's phenomenon (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=288) | Nintedanib (N=288)
Abdominal pain (Gastrointestinal disorders) | 21 | 36
Abdominal pain upper (Gastrointestinal disorders) | 15 | 21
Constipation (Gastrointestinal disorders) | 19 | 15
Diarrhoea (Gastrointestinal disorders) | 92 | 218
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 26 | 20
Nausea (Gastrointestinal disorders) | 41 | 96
Vomiting (Gastrointestinal disorders) | 31 | 78
Fatigue (General disorders) | 21 | 33
Pyrexia (General disorders) | 13 | 20
Bronchitis (Infections and infestations) | 27 | 22
Influenza (Infections and infestations) | 15 | 16
Nasopharyngitis (Infections and infestations) | 56 | 43
Respiratory tract infection (Infections and infestations) | 16 | 10
Upper respiratory tract infection (Infections and infestations) | 43 | 39
Urinary tract infection (Infections and infestations) | 28 | 28
Alanine aminotransferase increased (Investigations) | 4 | 22
Aspartate aminotransferase increased (Investigations) | 1 | 16
Gamma-glutamyltransferase increased (Investigations) | 4 | 19
Weight decreased (Investigations) | 15 | 39
Decreased appetite (Metabolism and nutrition disorders) | 14 | 28
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 15
Dizziness (Nervous system disorders) | 15 | 19
Headache (Nervous system disorders) | 28 | 34
Cough (Respiratory, thoracic and mediastinal disorders) | 62 | 41
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 | 23
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 | 8
Skin ulcer (Skin and subcutaneous tissue disorders) | 54 | 56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT02597933/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/33/NCT02597933/SAP_001.pdf